CLINICAL TRIAL: NCT05018741
Title: Prognostic Factors After Liver Transplantation
Status: Completed | Type: Observational
Sponsor: Changhua Christian Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 191244
Record Dates: First submitted 2021-08-22; First posted 2021-08-24 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Liver Diseases; Liver Transplant; Complications
Keywords: liver transplantation; chronic liver disease; viral hepatitis; alcoholic liver disease
MeSH Terms: conditions — Liver Diseases; Liver Diseases, Alcoholic | interventions — Liver Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Liver transplant
  Interventions: Procedure: liver transplantation

INTERVENTIONS:
Procedure: liver transplantation — liver transplantation for chronic liver disease or acute liver failure

SUMMARY:
The study retrospectively reviewed the medical records of patients who received adult liver transplantation in Changhua Christian hospital from 2002 to 2019. We collected their personal data about liver disease, laboratory data about liver function, pre-transplant evaluation and post-transplant outcome. We investigate what prognostic factors may contribute a good survival outcome, and improve our clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* patients who received adult liver transplantation in Changhua Christian hospital from 2002 to 2019

Exclusion Criteria:

* patients who did not have suitable donor for liver transplantation

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with acute liver failure or chronic liver disease due to different etiologies received liver transplantation
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2002-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
number of participants with morbidity and mortality after surgery | upto one month after surgery
  post-operative complications which requiring interventions, related to organ failure and hospital mortality

SECONDARY OUTCOMES:
long-term survival rate | upto 5 years after surgery
  1,5 year survival rate

CONTACTS AND LOCATIONS:
Overall Officials: Yao-Li Chen, Study Chair — Department of General Surgery, Changhua Christian Hospital, Changhua, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee SG, Hwang S, Moon DB, Ahn CS, Kim KH, Sung KB, Ko GY, Park KM, Ha TY, Song GW. Expanded indication criteria of living donor liver transplantation for hepatocellular carcinoma at one large-volume center. Liver Transpl. 2008 Jul;14(7):935-45. doi: 10.1002/lt.21445. PMID 18581465
- [Background] Chang Y, Cho Y, Lee JH, Lee YB, Cho EJ, Yu SJ, Sinn DH, Kim BH, Kim SH, Yi NJ, Lee KW, Kim JM, Park JW, Kim YJ, Yoon JH, Joh JW, Suh KS. Comparison of Models for Tumor Recurrence after Liver Transplantation for the Patients with Hepatocellular Carcinoma: A Multicenter Long-Term Follow-Up Study. Cancers (Basel). 2019 Sep 3;11(9):1295. doi: 10.3390/cancers11091295. PMID 31484287
- [Result] Mazzaferro V, Llovet JM, Miceli R, Bhoori S, Schiavo M, Mariani L, Camerini T, Roayaie S, Schwartz ME, Grazi GL, Adam R, Neuhaus P, Salizzoni M, Bruix J, Forner A, De Carlis L, Cillo U, Burroughs AK, Troisi R, Rossi M, Gerunda GE, Lerut J, Belghiti J, Boin I, Gugenheim J, Rochling F, Van Hoek B, Majno P; Metroticket Investigator Study Group. Predicting survival after liver transplantation in patients with hepatocellular carcinoma beyond the Milan criteria: a retrospective, exploratory analysis. Lancet Oncol. 2009 Jan;10(1):35-43. doi: 10.1016/S1470-2045(08)70284-5. Epub 2008 Dec 4. PMID 19058754